CLINICAL TRIAL: NCT00234182
Title: Postoperative Adjuvant Therapy With Recombinant Interferon-Alpha Following Curative Resection of Hepatocellular Carcinoma: a Randomized Controlled Trial
Brief Title: Postoperative Adjuvant Therapy With Recombinant Interferon-Alpha Following Curative Resection of HCC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC 1018-98
Record Dates: First submitted 2005-10-05; First posted 2005-10-06 (Estimated); Last update posted 2005-12-01 (Estimated); Status verified 2005-10

CONDITIONS: Hepatocellular Carcinoma
Keywords: liver cancer; hepatectomy; survival; recurrence
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms; Recurrence | interventions — Introns

INTERVENTIONS:
Drug: Interferon alpha-2b

SUMMARY:
We conducted a randomized controlled trial of adjuvant interferon therapy in patients with predominantly hepatitis B-related hepatocellular carcinoma (HCC) to investigate whether the prognosis after hepatic resection could be improved. Since February 1999, patients with no residual disease after hepatic resection for HCC were randomly assigned with stratification by pTNM stage to receive no treatment (control group), interferon alpha-2b 10 MIU/m2 (IFN-I group) or 30 MIU/m2 (IFN-II group) thrice weekly for 16 weeks. Enrollment to the IFN-II group was terminated from January 2000 because adverse effects resulted in treatment discontinuation in the first 6 patients. By June 2002, 40 patients each had been enrolled into the control group and IFN-I group. The baseline clinical, laboratory and tumor characteristics of both groups were comparable. The 1- and 5-year survival rates were 85% and 61%, respectively for the control group and 97% and 79%, respectively for the IFN-I group (P=0.137). After adjusting for the confounding prognostic factors in a Cox model, the relative risk of death for interferon treatment was 0.42 (95% CI 0.17 - 1.05; P=0.063). Exploratory subset analysis showed that adjuvant interferon had no survival benefit for pTNM stage I/II tumor (5-year survival 90% in both groups; P=0.917) but prevented early recurrence and improved the 5-year survival of patients with stage III/IVA tumor from 24% to 68% (P=0.038). In conclusion, in a group of patients with predominantly hepatitis B-related HCC, adjuvant interferon therapy prevented early recurrence and improved survival in those with pTNM stage III/IVA tumors.

DETAILED DESCRIPTION:
1. Background

   Hepatocellular carcinoma (HCC) is the second commonest cause of cancer death in Hong Kong and the majority are hepatitis B related. Hepatic resection has remained the only therapeutic option that can offer these patients a chance of long-term survival. Although the safety of hepatectomy has improved, postoperative recurrences are frequent. Depending on the size of the primary tumors, recent reports from Japan, France and Hong Kong1 showed that the postoperative recurrence rate was 20 to 64% at one year and 57 to 81% at 3 years.

   While the hepatic remnant is the predominant site of recurrence, involvement of extrahepatic organs was not infrequent. There are three possible mechanisms for the development of recurrent disease:

   i) residual tumor cells due to an inadequate resection margin ii) subclinical metastasis that occurs before or during hepatic resection iii) metachronous multicentric hepatocarcinogenesis which may be related to the underlying necroinflammation of chronic active hepatitis and oncogenic activities of hepatitis viruses.

   The surgeon's attempt to prevent recurrence by more extensive resection is prohibited by the need to preserve hepatic function. Futhermore, even a major hepatic resection cannot guarantee freedom from recurrence since metachronous multicentric tumors can develop in the entire liver. Theorectically, total hepatectomy and liver transplantation removes both the subclinical metastases in the liver and prevent metachronous lesions. Unfortunately, with immunosuppressive therapy, recurrences are frequent and tumors grow more rapidly, thus, illustrating the importance of the host immune surveillance in preventing the development of recurrence.

   The use of postoperative regional and systemic chemotherapy has been reported. Although retrospective studies have shown encouraging results, there are only limited number of prospective trials. The favourable result of the use of oral 1-hexylcarbomyl-5-fluorouracil in a multi-center trial as reported by Yamamoto and colleagues was questionable since treatment was suspended due to side-effects in 44% of the patients. Our single-center prospective randomised study performed at Queen Mary Hospital (QMH) using a combination of transarterial chemoembolisation and systemic epirubicin showed a higher extrahepatic recurrence rate and worse outcome with the use of adjuvant chemotherapy. The reasons for the failure of adjuvant chemotherapy include:

   i) HCC is slow-growing and hence cytotoxic drug resistant. ii) the associated liver cirrhosis limits the maximum tolerated intensity of chemotherapy iii) the anticancer agents may adversely affect the host immunity
2. Interferon alpha-2b

   Interferon alpha-2b is a recombinant form of human interferon. Interferons are cytokines possessing anti-viral, anti-proliferative and immunodulatory effects. Interferon may halt the replication of both hepatitis B and hepatitis C virus, thus, reducing the severity of the chronic active hepatitis. The histologic activity of chronic active hepatitis is an important risk factor for recurrence related to metachronous multicentric hepatocarcinogenesis and the use of interferon has been shown to reduce the incidence of HCC in patients with cirrhosis due to hepatitis C and possibly hepatitis B.

   Interferon has a powerful anti-proliferative effect on hepatoma cell-line PLC/PRF/5 in a dose-dependent manner both in-vitro and in-vivo. The use of interferon has been applied to patients with inoperable HCC with a tumour regression rate and survival rate superior to that of placebo-control or chemotherapeutic agents such as doxorubicin.

   Peripheral blood mononuclear cells from patients with HCC have considerably reduced cytotoxicity against hepatoma cell lines. Interferon has been shown to normalise the T-lymphocyte subpopullation and enhance the cytotoxic activity against an HBsAg-producing hepatoma cell line in-vitro.
3. Interferon adverse effects

   Interferon alpha-2b is registered for treatment of HCC and chronic hepatitis B in Hong Kong. In patients with unresectable HCC, interferon has a much lower incidence of fatal side-effects when compared to doxorubicin. Most patients experience flu-like symptoms including fever, headache, fatigue and myalgia which usually subside spontaneously with continuation of treatment. Less common but more serious adverse effects include alopecia, leukopenia, thrombocytopenia, depression, irritability, and mental deterioration. The adverse effects are dose-dependent and the majority are reversible with a reduction in dosage. The use of high-dose interferon has been well-tolerated in clinical trials involving patients with unresectable HCC.
4. Rationale

Interferon has anti-viral, anti-proliferative and immunodulatory activities. It has been used clinically in the treatment of unresectable HCC as well as viral hepatitis B and C. It can potentially reduce the incidence of recurrence due to residual tumour cells or metachronous multicentric disease in patients after resection for HCC.

ELIGIBILITY:
Inclusion Criteria:

All patients who undergo a curvative hepatic resection for HCC at the Department of Surgery, Queen Mary Hospital are included. The criteria for curative resection include all of the following :

i) Complete extirpation of disease as demonstrated by intraoperative ultrasonography during surgery ii) Histologic evidence of a clear resection margin iii) No evidence of residual disease in the liver remnant as demonstrated by spiral contrast-enhanced CT scan one month after surgery

Exclusion Criteria:

i) patient refusal ii) age > 75 years old iii) hospital mortality iv) disease previously treated by regional or systemic chemotherapy, hormonal therapy or immunotherapy v) poor hepatic function:

1. presence of hepatic encephalopathy
2. presence of ascites not controlled by diuretics
3. history of variceal bleeding within last 3 months
4. total serum bilirubin > 50 umol/L
5. serum albumin < 30 g/L
6. prothrombin time prolonged for > 4 seconds vi) poor renal function with serum creatinine > 180mol/L vii) Absolute neutrophil count < 1.5 x 109/L viii) Platelet count < 75 x 109/L ix) poor performance status with European Cooperative Oncology Group (ECOG) scale grade III or IV

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84
Dates: Start 2000-01; Study Completion 2004-12

PRIMARY OUTCOMES:
Occurrence of recurrent disease

SECONDARY OUTCOMES:
Death of the patient

CONTACTS AND LOCATIONS:
Overall Officials: Chung Mau Lo, MS, Principal Investigator — Department of Surgery, The University of Hong Kong